CLINICAL TRIAL: NCT04558411
Title: Pilot Study of a Brief, Scaleable Intervention for COVID-19 Mental Health Sequelae in College Students
Brief Title: Brief, Scaleable Intervention for Coronavirus (COVID-19) Mental Health Sequelae in College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Shireen L. Rizvi, PhD, ABPP, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2020002008
Record Dates: First submitted 2020-09-20; First posted 2020-09-22 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Emotional Regulation; Affect
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (assessment only) (No Intervention): This group will receive assessments only.
- Assessment + Intervention Group (Experimental): This group will receive assessments and the 14 brief intervention videos.
  Interventions: Behavioral: Dialectical Behavioral Therapy (DBT) Skills

INTERVENTIONS:
Behavioral: Dialectical Behavioral Therapy (DBT) Skills — 14 brief videos that teach DBT skills.
  Arms: Assessment + Intervention Group

SUMMARY:
The major aim of this pilot study is to evaluate a brief coping skills intervention for college students, based on an evidence-based treatment and delivered remotely via 14 short daily videos. Participants will be 150 Rutgers undergraduates who are enrolled in Fall 2020. Participants in the experimental group (n=100) will receive 4 daily smartphone surveys assessing stress, affect, and other related factors for two weeks before, during, and after the 2-week coping skills intervention. Participants in the control group (n=50) will receive assessments over the same time period with no skills intervention. Both groups will be assessed weekly throughout the Fall semester to monitor the transition to the new semester and longer-term impact of the intervention. The control condition participants will have access to the skills videos at the end of the study.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older
* Matriculated at Rutgers during Fall of 2020 (on campus and/or remote)
* Currently residing in the United States
* Willingness to follow study requirements, as evidenced by an ability to provide written informed consent and read, understand, and complete the study procedures
* iOS and Android smartphone compatible with MetricWire

Exclusion Criteria

* Non-English speaking
* Unable to understand or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Distress | Six week daily monitoring period
  Distress, as assessed via smartphone Ecological Momentary Assessment (EMA), 0 through 10 scale, 10 equals more distress.
Emotion regulation | Six week daily monitoring period
  Assessed with the Difficulties in Emotion Regulation Scale (DERS); scores range from 36-180, higher scores equal more distress
Distress (within-person change) | Six week daily monitoring period
  Assessed via EMA in the experimental group, 0 through 10 scale, 10 equals more distress.

SECONDARY OUTCOMES:
Maintenance of improvement in emotion regulation | Six week post-daily monitoring period
  Assessed with the Difficulties in Emotion Regulation Scale (DERS), scores range from 36-180, higher scores equal more distress

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers, The State University of New Jersey, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share data after the publication of primary manuscripts.
Supporting Information: Study Protocol, Analytic Code
Time Frame: We will share data after the publication of primary manuscripts.